CLINICAL TRIAL: NCT01345708
Title: A Single-Arm Pilot Study With Low-Dose Rituximab Plus Standard Oral Prednisone In Idiopathic Autoimmune Hemolytic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: University Hospital, Udine, Italy (Other)
Responsible Party: Wilma Barcellini, MD, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eudra CT 2008-006713-25
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Autoimmune Hemolytic Disease (Cold Type) (Warm Type)
Keywords: Low dose rituximab; WAIHA; CHD
MeSH Terms: interventions — Prednisone; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: prednisone, low dose rituximab — Patients with "warm" AIHA will receive:
  Rituximab 100 mg i.v.weekly (fixed dose irrespective of body surface area) for 4 consecutive weeks (days +7, +14, +21, +28), and prednisone 1 mg/kg/die p.o. days from day +1 to day +30, followed by tapering (10 mg/week until 0.5/mg/kg/die, then 5 mg/week until stop)
  Patients with CHD will receive:
  Rituximab 100 mg i.v.weekly (fixed dose irrespective of body surface area) for 4 consecutive weeks (days +7, +14, +21, +28)

SUMMARY:
The aim of this prospective study was to evaluate the activity, safety and the duration of the response of low dose rituximab associated with standard oral prednisone as first line therapy in newly diagnosed warm autoimmune hemolytic anemia and cold hemagglutinin disease, and as second line therapy in warm autoimmune hemolytic anemia relapsed after standard oral prednisone. Further aim was to correlate the clinical response to biological parameters (cytokine and anti-erythrocyte antibody production in cultures).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed "warm" or "cold" AIHA, defined by symptomatic anemia and positive DAT, in the absence of underlying lymphoproliferative, infectious or neoplastic disease (according to the single Center diagnostic criteria).
* Idiopathic "warm" or "cold" AIHA relapsed after first line treatment with oral prednisone.
* Aged >18 years
* ECOG performance status grade 0, 1 or 2
* No psychiatric illness that precludes understanding concepts of the trial or signing informed consent
* Patients who have provided written informed consent prior to study participation, with the understanding that the consent may be withdrawn by the patient at any time without prejudice.

Exclusion Criteria:

* Cell or humoral immunologic deficit (congenital or acquired)
* Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent
* Active bacterial, viral, or fungal infection requiring systemic therapy HIV or HbsAg positive (with HBV-DNA+) or HCV-Ab positive (with HCV-RNA+) patients
* History of malignancies within 3 years prior to study entry
* Concomitant immunosuppressive or cytotoxic treatment
* Positive pregnancy test. Lactation.
* The presence of associated organ-specific autoimmune diseases do not constitute exclusion criteria. Previous splenectomy does not constitute exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
overall response | month +2
  Response will be evaluated at each clinic visit. Complete response (CR) will be defined as Hb increase >2 g/dL and Hb > 12 g/dL, normalization of all haemolytic markers and no transfusion requirement;Partial response (PR) will be defined as Hb increase >2 g/dL and Hb 10-12 g/dL, and 50% reduction of transfusion. In the remaining cases there is no response.

SECONDARY OUTCOMES:
Sustained response (SR) | month +6, month +12
  Sustained response (SR) was defined as Hb > 10 g/dL at month +6 and +12, in the absence of any treatment.

CONTACTS AND LOCATIONS:
Overall Officials: PierMannuccio Mannucci, MD, Study Director — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Via F. Sforza 28 20122, Milano.
Locations (2):
- Italy (2):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Wilma Barcellini MD, UO Ematologia 2, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan

REFERENCES:
- [Background] Provan D, Butler T, Evangelista ML, Amadori S, Newland AC, Stasi R. Activity and safety profile of low-dose rituximab for the treatment of autoimmune cytopenias in adults. Haematologica. 2007 Dec;92(12):1695-8. doi: 10.3324/haematol.11709. PMID 18055995
- [Background] Zaja F, Vianelli N, Volpetti S, Battista ML, Defina M, Palmieri S, Bocchia M, Medeot M, De Luca S, Ferrara F, Isola M, Baccarani M, Fanin R. Low-dose rituximab in adult patients with primary immune thrombocytopenia. Eur J Haematol. 2010 Oct;85(4):329-34. doi: 10.1111/j.1600-0609.2010.01486.x. Epub 2010 Jul 28. PMID 20546023
- [Background] Gomez-Almaguer D, Solano-Genesta M, Tarin-Arzaga L, Herrera-Garza JL, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Jaime-Perez JC. Low-dose rituximab and alemtuzumab combination therapy for patients with steroid-refractory autoimmune cytopenias. Blood. 2010 Dec 2;116(23):4783-5. doi: 10.1182/blood-2010-06-291831. Epub 2010 Sep 14. PMID 20841509
- [Derived] Barcellini W, Zaja F, Zaninoni A, Imperiali FG, Battista ML, Di Bona E, Fattizzo B, Consonni D, Cortelezzi A, Fanin R, Zanella A. Low-dose rituximab in adult patients with idiopathic autoimmune hemolytic anemia: clinical efficacy and biologic studies. Blood. 2012 Apr 19;119(16):3691-7. doi: 10.1182/blood-2011-06-363556. Epub 2012 Jan 20. PMID 22267606